CLINICAL TRIAL: NCT06253650
Title: Adjuvant TRastuzumab Deruxtecan Plus Fluoropyrimidine Versus Standard Chemotherapy In HER2-positive Gastric or Gastroesophageal Cancer Patients With Persistence of miNImal Residual Disease in Liquid Biopsy After Pre-operative chemoTherapy and Radical surgerY
Brief Title: Adjuvant TRastuzumab Deruxtecan for HER2-positive Gastroesophageal Cancer With Persistence of miNImal Residual Disease
Acronym: TRINITY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506662-31-00
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; HER2-positive Gastric Cancer
Keywords: Trastuzumab-Deruxtecan; Gastric Cancer; HER2-positive Gastric Cancer; Liquid biopsy; Minimal residual disease
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): treatment with T-DXd (6.4 mg/kg intravenous every 3 weeks) plus capecitabine (1000 mg/sqm BID orally on days 1-14 every 3 weeks) or 5-fluorouracil (600 mg/m2/day continuous intravenous infusion on days 1-5 every 3 weeks) as per Investigator's choice for 6 cycles.
  Interventions: Drug: Experimental
- Control (Active Comparator): treatment with post-operative FLOT for 4 cycles as per standard of care and using the doses previously adopted in the last cycle of the preoperative phase, i.e. 5-fluorouracil (2600 mg/m2 continuous intravenous infusion day 1 for 24 hours every 2 weeks), leucovorin (200 mg/m2 intravenous infusion on day 1 every 2 weeks), oxaliplatin 85 mg/m2 (intravenous infusion on day 1 every 2 weeks) and docetaxel (50 mg/m2 intravenous infusion on day 1 every 2 weeks).
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Experimental — 6 cycles of: T-DXd at the dose of 6.4 mg/kg intravenous every 3 weeks plus capecitabine 1000 mg/sqm BID orally on days 1-14 every 3 weeks or 5-fluorouracil 600 mg/m2/day continuous intravenous infusion on days 1-5 every 3 weeks as per Investigator's choice
  Arms: Experimental
Drug: Control — 4 cycles of: 5-fluorouracil 2600 mg/m2 continuous intravenous infusion day 1 for 24 hours every 2 weeks, leucovorin 200 mg/m2 intravenous infusion on day 1 every 2 weeks, oxaliplatin 85 mg/m2 intravenous infusion on day 1 every 2 weeks, and docetaxel 50 mg/m2 intravenous infusion on day 1 every 2 weeks.
  Arms: Control

SUMMARY:
TRINITY is designed as a multicentre, randomized, open-label, interventional phase II study aimed at investigating the activity, efficacy and safety of trastuzumab-deruxtecan (T-DXd) plus capecitabine/5-fluorouracil as a post-operative treatment in localized/locally advanced gastric or gastroesophageal junction cancer (GC/GEJC)/esophageal adenocarcinoma patients with HER2 overexpression/amplification and positive post-operative ctDNA after pre-operative 5-fluorouracil plus leucovorin, oxaliplatin, and docetaxel (FLOT) regimen followed by radical surgery.

DETAILED DESCRIPTION:
Patients affected by localized/locally advanced GC/GEJC (Siewert I-II-III)/esophageal adenocarcinoma eligible for peri-operative chemotherapy and radical surgery and deemed fit enough to receive the standard treatment with the triplet FLOT (5-fluorouracil, oxaliplatin and docetaxel) will be evaluated for the enrollment into the observational phase of the study during the standard pre-operative therapeutic management according to the best clinical practice and local guidelines at their Centre.

OBSERVATIONAL PHASE The observational phase will include patients with localized/locally advanced HER2-positive GC/GEJC (Siewert I-II-III)/esophageal adenocarcinoma eligible for standard pre-operative chemotherapy with FLOT for 4 cycles and radical surgery. Patients will undergo an exploratory liquid biopsy (LB) to be centrally collected at baseline, i.e. during the baseline disease staging as per standard clinical practice and prior to the start of the pre-operative FLOT treatment, and a second exploratory LB to be centrally collected at the end of the pre-operative FLOT treatment before the standard surgery. Then, a third mandatory exploratory LB will be collected at 2-6 weeks after surgery and, during the same timepoint, the interventional liquid biopsy will be collected and centrally analyzed with the SignateraTM CE-marked assay as pre-screening test ® in order to determine whether post-operative ctDNA is positive or negative (LB#1: interventional for the potential enrollment in the TRINITY study). Patients will be permitted to be enrolled in the observational phase even after the start of pre-operative FLOT or even after surgery, the lack of availability of one or both pre-surgical exploratory LBs will not preclude the enrolment in the interventional study and postoperative SignateraTM will be offered as prescreening assay.

Patients eligible for the interventional TRINITY study will be those who underwent surgery after the completion of the standard FLOT pre-operative treatment, with locally-confirmed HER2 positive status both on archival pre-treatment tumor biopsy and on post-treatment surgical sample and with detected post-operative ctDNA at LB#1.

In any case of non-eligibility for the interventional study for not fulfilling the molecular pre-screening algorithm, patients will continue the standard treatment as per clinical practice with post-operative FLOT for 4 cycles and standard follow up. In this case, patients with prescreening failure will continue to be followed-up in the frame of the observational phase of the study with the collection of serial LBs at specific timepoints at 3, 6 and 12 months from the date of pre-screening failure (date of results of LB#1), respectively, and then in concomitance with follow-up visits scheduled as per standard clinical practice.

INTERVENTIONAL TRINITY STUDY Patients deemed eligible for the Screening in the interventional TRINITY trial will be screened from 2 and 12 weeks after the date of surgery, in order to start the post-operative treatment no later than 12 weeks after surgery, and will undergo all the screening tests comprising a CT scan including high resolution thorax-abdomen CT scan and echocardiography.

Patients fulfilling all the eligibility criteria for the trial will be randomized according to a 1:1 basis to the experimental treatment with T-DXd at the dose of 6.4 mg/kg intravenous every 3 weeks plus either capecitabine 1000 mg/sqm BID orally on days 1-14 or 5-fluorouracil 600 mg/sqm continuous intravenous infusion on days 1-5, as per Investigator's choice, every 3 weeks for 6 cycles versus the control treatment arm with post-operative FLOT with standard dose and schedule and at the same dose used during the last pre-operative cycle, for 4 cycles.

At 3, 6 and 12 months after randomization, additional exploratory LBs will be collected and at 12 months after randomization also the interventional LB#2 will be collected and centrally analysed to detect ctDNA and to assess the occurrence of ctDNA clearance in both arms as per study primary endpoint.

After randomization, patients will undergo a thorax-abdomen CT scan every 3 months for 1 year to monitor the occurrence of clinical disease relapse. In case of disease relapse before the 12-month post-randomization time-point, the interventional LB#2 will not be performed. After 12 months post-randomization, exploratory LBs will be performed longitudinally during follow-up as per standard clinical practice. Importantly, exploratory LB will be always collected at the time of disease relapse.

This study will pre-screen approximately 600 patients, in order to include about 100 patients in the observational phase and enrol a total number of 46 patients in the interventional study, across 20 Italian Centres in the frame of the GONO network.

ELIGIBILITY:
Inclusion Criteria of the Interventional TRINITY study:

1. Written informed consent and any locally required authorization (such as the European Union [EU] Data Privacy Directive) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Compliance with all the study procedures and treatments. Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating Centre.
3. Age ≥ 18 years old.
4. Eastern Cooperative Oncology group (ECOG) Performance Status 0-1.
5. Life expectancy of at least 12 weeks.
6. Resected gastric or gastroesophageal junction (Siewert I-II-III) cancer/esophageal adenocarcinoma, after the completion of pre-operative chemotherapy with FLOT, as per standard clinical practice.
7. Absence of distant metastases as defined by post-operative radiological assessments (contrast-enhanced CT scan of the thorax and abdomen or, in case of contraindications, non-contrast-enhanced chest CT scan and abdomen Magnetic Resonance Imaging)
8. Presence of locally determined HER2 overexpression/amplification on the post-treatment surgical tissue specimen defined as IHC 3+ or 2+/ISH amplified.
9. Positivity of the post-operative liquid biopsy, performed 2-6 weeks after the radical surgery.
10. LVEF ≥ 50% within 28 days before randomization/enrolment.
11. Adequate bone marrow and organ function within 14 days before randomization/enrolment as described below:

    1. Neutrophil count ≥ 1.5 x 10^3/μL
    2. Platelet count ≥ 100 x 10^6/μL
    3. Haemoglobin ≥ 9 g/dL
    4. Total bilirubin lower than 1.5 time the upper-normal limits (ULN) of the Institutional normal values
    5. AST (SGOT) and/or ALT (SGPT) <3 x ULN
    6. serum albumin ≥ 2.5 g/dL
    7. Creatinine clearance (calculated according to Cockroft and Gault) > 60 mL/min
    8. International normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN
12. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of IMP. Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
13. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, from the time of screening and must agree to continue using such precautions for 7 months after the last dose of IMP. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
14. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP for T-DXd while 6 months for docetaxel and oxaliplatin. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of randomisation/enrolment, throughout the study and for 4 months after the last dose of IMP for T-DXd while 6 months for docetaxel and oxaliplatin. Preservation of sperm should be considered prior to enrollment in this study.
15. Female subjects must not donate, or retrieve for their own use, ova from the time of randomization/enrolmentand throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.

Exclusion Criteria of the Interventional TRINITY study:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Participation in another clinical study with an investigational product during the last 12 months
3. Signs of distant metastases at any site.
4. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, renal disease, neurological disease or peripheral neuropathy, serious chronic gastrointestinal conditions associated with diarrhea, or substance abuse or any other medical or psychiatric illness/social situations that in the opinion of the investigator would limit compliance with study requirement, interfere with the subject's participation in the clinical study, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent or interfere with the evaluation of the clinical study results.
5. Patients with a medical history of myocardial infarction (MI) within 6 months before randomization/enrolment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI.
6. Corrected QT interval (QTcF) prolongation to > 470 msec (females) or >450 msec (males) based on average of the screening triplicate12-lead ECG.
7. History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
8. Lung criteria:

   * Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
   * Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
   * Prior pneumonectomy (complete)
9. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
10. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection not under adequate disease control (that is defined as the presence of all the following conditions: receiving stable regimen of highly active anti-retroviral therapy for at least 4 weeks prior to study enrollment, CD4+ count above 250 cells/μL, undetectable viral load on standard polymerase chain reaction-based tests, absence of any HIV-related opportunistic infections for at least 4 weeks prior to study enrollment and no requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections), or active hepatitis B or C infection (HBsAg, anti-HBs, anti-HBc, anti-HCV). Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients who are anti-HBc positive and HBsAg negative or patients with HBsAg positive have to dose HBV-DNA. If HBV DNA is undetectable (<10UL/ml or under the limit of detection per local lab standard) are considered as HBV negative. Subjects should be tested for HIV prior to randomization/enrollment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
11. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of T-DXd. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP.
12. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline. Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to [randomization/enrollment/Cycle 1 Day 1] and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as: chemotherapy-induced neuropathy and fatigue.
13. Known allergy or hypersensitivity to study treatment or any of the study drug excipients.
14. History of severe hypersensitivity reactions to other monoclonal antibodies.
15. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.
16. Multiple primary malignancies within 3 years, except for

    * adequately resected non-melanoma skin cancer
    * curatively treated in-situ disease
    * other solid tumors curatively treated
17. A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).
18. LVEF< 50% within 28 days before enrolment.
19. Prior treatment with an anti-HER2 agent.
20. Absence of locally determined HER2 overexpression/amplification on the surgical specimen defined as IHC 0 or 1+ or 2+/ISH not amplified.
21. Negativity of ctDNA at the post-operative liquid biopsy.

21. Known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency based on local laboratory testing before the start of pre-operative FLOT regimen. Confirmation of the assessment of DPD status before the start of pre-operative FLOT in the patient's records should be provided before the enrollment in the interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance (negative ctDNA status) at 1 year | 1 year
  The clearance of ctDNA in T-DXd plus capecitabine/5-fluorouracil arm versus standard FLOT continuation at 1 year from randomization.

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  time from the randomization in the study to the occurrence of disease relapse (local and/or distant), second GC/GEJC primary, or death from any cause
Overall survival | 3 years
  time from the randomization in the study to the occurrence of death.
Metastases-free survival | 3 years
  time from the randomization in the study to the first evidence of metastases according to the radiological and clinical assessments detailed in the procedures or death from any cause.
Quality of life - PRO EORTC-QLQ-C30 | during adjuvant treatment phase
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-C30 For questions 1-28 of EORTC QLQ-C30 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit")and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. For the questions 29 and 30 of EORTC QLQ-C30 a 7-points scale is used. It scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Quality of life - EORTC QLQ-STO22 | during adjuvant treatment phase
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-STO22.
  For questions 31-52 of EORTC QLQ-STO22 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
Quality of life - PRO EuroQol EQ-5D-5L | during adjuvant treatment phase
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EuroQol EQ-5D-5L. The EQ-5D-5L uses for first 5 questions qualitative multiple choice answers with NO SCALE. For the last questions, a score from 0 to 100 indicates from the worst to the best outcome.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months
  incidence of adverse events during the treatment and follow-up phases, assessed according to CTCAE v5.0.

OTHER OUTCOMES:
Translational analyses | 3 years
  To conduct exploratory translational analyses aimed at identifying which subgroup of patients may derive the highest benefit from a post-operative targeted treatment with T-DXd as compared to FLOT continuation after pre-operative FLOT and radical surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS - Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The trial results concerning the primary, secondary and exploratory outcomes will be published according to the standard guidelines. IPD could eventually be requested to the Sponsor and Principal Investigator, who will carefully evaluate the formal and motivated request.

REFERENCES:
- [Derived] Nasca V, Bergamo F, Foltran L, Antonuzzo L, Bencardino K, Dell'Aquila E, Corallo S, Spallanzani A, Brunetti O, Spada D, Tamberi S, Cella CA, Avallone A, Fornaro L, Di Donato S, Strippoli A, Puccini A, Tamburini E, Palermo F, Morano F, Pietrantonio F, Raimondi A. Adjuvant TRastuzumab deruxtecan plus fluoropyrimidine versus standard chemotherapy in HER2-positive gastric or gastroesophageal cancer patients with persistence of minimal residual disease in liquid biopsy after pre-operative chemotherapy and radical surgery: the multicentre, phase II randomized TRINITY trial. BMC Cancer. 2025 Apr 8;25(1):633. doi: 10.1186/s12885-025-14063-6. PMID 40200187